CLINICAL TRIAL: NCT04111003
Title: Fiber-reinforced Composite Core Filling in the Restoration of Endodontically Treated Molars - a Clinical Study
Acronym: sFRCendocr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: GC Europe (Industry); City of Turku (Other Government)
Responsible Party: Principal Investigator, Johanna Tanner, Associate professor, Department of Prosthetic Dentistry and Stomatognathic Physiology, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20341 601350
Record Dates: First submitted 2017-10-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Dental Materials; Tooth, Nonvital
Keywords: fiber-reinforced composite
MeSH Terms: conditions — Tooth, Nonvital | interventions — Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFRC direct filling (Experimental): Restoration of endodontically treated tooth Endodontically treated molars are restored with direct composite restorations, using a short-FRC base filling.
  Interventions: Procedure: local anesthesia; Procedure: Tooth restored using SFRC filling
- CEREC endocrown (Active Comparator): Restoration of endodontically treated tooth Endodontically treated molars are restored with indirect ceramic CAD/CAM restorations.
  Interventions: Procedure: local anesthesia; Procedure: Tooth restored using Ceramic indirect endocrown

INTERVENTIONS:
Procedure: local anesthesia — administering local anesthesia in the region of the planned restorative procedure
Procedure: Tooth restored using SFRC filling — Restoration of an endodontivally treated molar using a shor-fiber base filling and veneering composite
  Arms: SFRC direct filling
Procedure: Tooth restored using Ceramic indirect endocrown — Restoration of an endodontically treated molar using a ceramic indirect restoration
  Arms: CEREC endocrown

SUMMARY:
A short fiber reinforced composite base filling material has been shown to improve the strength of a direct composite filling significantly. It prevents fracture propagation and reduces shrinkage strain. These features are needed especially in endodontically treated molars, as root-canal treated teeth are structurally compromised and their restoration is associated with technical failures such as debonding and vertical root fractures.

Application on this core fiber-reinforced composite (FRC) material is simplified when compared to post and core techniques commonly used to restore endodontically treated teeth. Clinically, the use of core FRC offers a cost-effective way to restore endodontically treated molars without root canal involvement.

The purpose of this study is to compare the clinical performance of endodontically treated molars restored with either direct composite restorations with a FRC substructure, or with indirect full-ceramic onlay restorations, i.e. endo-crowns.

DETAILED DESCRIPTION:
INTRODUCTION

Composite resins are routinely used for restoring vital and non-vital posterior teeth by most practitioners in Finland. Various clinical studies have found that the three main reasons for failure of direct composite fillings are secondary caries, wear and fracture of composite resin especially at molar region (1, 2, 3). Non-vital (endodontically treated) teeth are structurally compromised and their restoration is associated with technical failures such as debonding and vertical root fractures (4). Techniques, like root canal post insertion, that are used to overcome these problems, are time consuming and may even further increase the risk for root fractures.

This study is a continuum on material development conducted at the the Department of Prosthetic Dentistry, Biomaterials Science and Turku Clinical Biomaterials Centre - TCBC, University of Turku, in collaboration with TEKES (Technology Development Center of Finland) and StickTech (Turku, Finland). The data obtained has shown that, the use of a bilayered structure consisting of a fiber-reinforced composite substructure (core FRC) combined with an upper layer of conventional restorative composite, increases the fracture load of a restoration significantly (5,6 and 7). This newly developed material has increased mechanical properties when compared to conventional materials, while maintaining its clinical applicability. Moreover, volumetric polymerization shrinkage of the core FRC is found to be lower than commercially available composites (<1.8% for the new FRC-material; 2.0% for a commercial composite Z250) (8). This may be expected to result in less marginal leakage and secondary caries in long term. With this backround a multidirectional short-fiber composite (everX, StickTech) has been introduced as a base material (FRC substructure) for large cavities in vital or non-vital teeth.

The investigators in vitro experiments have shown that the FRC substructure retains and significantly reinforces composite crowns in endodontically treated molars. Moreover, in case of failure, the presence of the FRC substructure seems to orient the fracture propagation and result in more easily restorable fractures. Application on the core FRC material is simplified when compared to post and core techniques commonly used to restore endodontically treated teeth. Clinically, the use of core FRC offers a cost-effective way to restore endodontically treated molars without root canal involvement. In a recently published clinical pilot study the investigators have reported successful 1 year results of this technique (9).

Ceramic onlay-restorations, so called "endo-crowns", are currently used to restore endodontically treated molars with similar indications (without root canal involvement). Case studies have reported good clinical results with this type of method (10). The use of an indirect technique (multiple patient visits), material and technical fabrication costs make this treatment modality, however, more costly and not in the reach of every patient.

.

AIM OF STUDY

The purpose of this study is to compare the clinical performance of endodontically treated molars restored with either direct composite restorations with a FRC subtructure, or with indirect full-ceramic onlay restorations, i.e. endo-crowns.

Specific study hypotheses are:

1. The five year survival of direct FRC restorations is equal to that of ceramic endo-crowns
2. Direct FRC restorations and ceramic endo-crowns perform equally with regard to

   1. marginal integrity
   2. fracture resistance
   3. occlusal wear
   4. secondary caries
3. Less bleeding on probing is present around ceramic restorations when compared to composite restorations
4. Less chair-side time is needed to restore a tooth with a direct FRC restoration than with a ceramic endo-crown

MATERIALS AND METHODS

The study will be carried out at the Institute of Dentistry of Turku University at Dentalia building (Lemminkäisenkatu 2, Turku). Subjects are enrolled among the patients of the undergraduate dental students (Dental teaching clinic, Turku city health care). Operators are experienced dental practitioners. Ethical committee approval was obtained (20.6.2006) form the Joint Commission on Ethics of the Turku University and The Turku University Hospital. A written informed concent will be obtained from all participants prior to their enrolment in the study.

Exclusion/inclusion is based on anamnestic data, clinical and radiographic examination. Exlusion criteria at patient level are known nocturnal bruxism, active periodontal disease and poor oral hygiene. Exclusion criteria at tooth level are: periapical pathosis, root canal filling >3 mm short from apex, vertical fracture observed in cavum dentin, more than 50% of cavity margin situated subgingivally, less than 2mm of coronal tooth tissue present and lack of occluding antagonist.

Alltogether 30 restorations, 15 direct composite restorations and 15 ceramic restorations, are made in endodontically treated posterior teeth (molars and premolars). Study teeth are randomly divided into two groups, the other receiving direct composite fillings and the other indirect ceramic fillings. In the composite group root canal orifices and the pulpal chamber is filled with the FRC substructure material forming a core restoration (everX, StickTech) and covered with an upperlayer of commercial restorative composite (Filtek Supreme 3M ESPE). In the ceramic group teeth are prepared for endo-crowns and optical impressions are made. CAD/CAM ceramic fillings are fabricated (CEREC, Dentsply Sirona) and subsequently cemented with resin cement at place. Special attention is payed to finishing and occlusal adjustment of the studied restorations.

Chair-side time consumed in the making of the studied restorations is recorded in order to determine the cost-effectiveness of the methods.

In addition to clinical examination, two to three visits per patient are required to fabricate the studied restorations. Impressions of the preparations are taken of all teeth to study the effect of remaining coronal tissue on the clinical survival.

Patients are recalled and restorations examined at yearly follow-up visits up to five years. The clinical appearance, marginal integrity, fracture resistance, occlusal wear and color stability as well as the condition of marginal periodontal tissues close to the studied materials are assessed.

X-rays at baseline, 2 and 5 year follow-up visits, are taken to determine the periapical status of the teeth and the intergrity of the restorations. Accordingly, impressions are taken and gypsum models casted to study the occlusal wear rate of the restorations.

STUDY TIMETABLE

Patient enrolling and examination, fall 2012 Clinical procedures, fabrication of restorations, 2012 - 2013 Follow-up examinations, 2013 - 2018 Analysing and reporting of the results, , 2018-2019

ELIGIBILITY:
Inclusion Criteria:

* need for a restoration in a endodontically treated upper of lower molar tooth
* adequate coronal tooth substance present for an adhesive restorative technique

Exclusion Criteria:

* propable sleep bruxism
* active periodontitis
* disability to performs oral hygiene measures
* periapical parodontitis in the study tooth
* low quality of root canal obturation
* fracture-line detected at cavity preparation
* no enamel present
* less than 2mm of coronal tissue present in average
* no opposing tooth

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2017-02-12 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Restoration failure detected at clinical follow-up examination | 5 years
  Observer scores the restoration having a fracture or detachment that requires remaking of the restoration.

SECONDARY OUTCOMES:
Restoration fracture detected at clinical follow-up examination | 5 years
  Observer scores the restoration having a fracture, which needs a repair
Restored tooth demonstrates with an endodontic complication needing removal of restoration or tooth. Clinical and radiographic examination requiered. | 5 years
  an endodontic infection requiring an endodontic retreatement or the loss of the tooth due to an endodontic infection
Observer scores the restoration having with dental caries at clinical follow-up investigation | 5 years
  Secondary dentinal caries, that requires restorative treatment, is observed adjacent to the restoration

CONTACTS AND LOCATIONS:
Overall Officials: Pekka K Vallittu, professor, Study Chair — University of Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarrett DC. Clinical challenges and the relevance of materials testing for posterior composite restorations. Dent Mater. 2005 Jan;21(1):9-20. doi: 10.1016/j.dental.2004.10.001. PMID 15680997
- [Background] van Dijken JW, Sunnegardh-Gronberg K. Fiber-reinforced packable resin composites in Class II cavities. J Dent. 2006 Nov;34(10):763-9. doi: 10.1016/j.jdent.2006.02.003. Epub 2006 Mar 31. PMID 16580114
- [Background] Manhart J. Direct composite restorations in posterior region: a case history using a nanohybrid composite. Dent Today. 2004 Nov;23(11):66, 68-70. No abstract available. PMID 15622879
- [Background] Torbjorner A, Karlsson S, Odman PA. Survival rate and failure characteristics for two post designs. J Prosthet Dent. 1995 May;73(5):439-44. doi: 10.1016/s0022-3913(05)80072-1. PMID 7658393
- [Background] Garoushi S, Lassila LV, Tezvergil A, Vallittu PK. Load bearing capacity of fibre-reinforced and particulate filler composite resin combination. J Dent. 2006 Mar;34(3):179-84. doi: 10.1016/j.jdent.2005.05.010. Epub 2005 Sep 8. PMID 16150524
- [Background] Garoushi SK, Lassila LV, Tezvergil A, Vallittu PK. Fiber-reinforced composite substructure: load-bearing capacity of an onlay restoration and flexural properties of the material. J Contemp Dent Pract. 2006 Sep 1;7(4):1-8. PMID 16957785
- [Background] Fennis WM, Kuijs RH, Kreulen CM, Verdonschot N, Creugers NH. Fatigue resistance of teeth restored with cuspal-coverage composite restorations. Int J Prosthodont. 2004 May-Jun;17(3):313-7. PMID 15237878
- [Background] Tezvergil A, Lassila LV, Vallittu PK. The effect of fiber orientation on the polymerization shrinkage strain of fiber-reinforced composites. Dent Mater. 2006 Jul;22(7):610-6. doi: 10.1016/j.dental.2005.05.017. Epub 2005 Oct 18. PMID 16239026
- [Background] Garoushi S, Tanner J, Vallittu P, Lassila L. Preliminary clinical evaluation of short fiber-reinforced composite resin in posterior teeth: 12-months report. Open Dent J. 2012;6:41-5. doi: 10.2174/1874210601206010041. Epub 2012 Jan 6. PMID 22408696
- [Background] van Dijken JW, Hasselrot L. A prospective 15-year evaluation of extensive dentin-enamel-bonded pressed ceramic coverages. Dent Mater. 2010 Sep;26(9):929-39. doi: 10.1016/j.dental.2010.05.008. Epub 2010 Jun 17. PMID 20691334